CLINICAL TRIAL: NCT01286818
Title: A Phase 1b Study of Irinotecan, Levofolinate, and 5-Fluorouracil (FOLFIRI) Plus Ramucirumab (IMC-1121B) Drug Product in Japanese Subjects With Metastatic Colorectal Carcinoma Progressive During or Following First-Line Combination Therapy With Bevacizumab, Oxaliplatin, and a Fluoropyrimidine
Brief Title: A Study of Irinotecan, Levofolinate, and 5-Fluorouracil (FOLFIRI) Plus Ramucirumab (IMC-1121B)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14223; CP12-1029 (Other: ImClone Systems); 14T-IE-JVBY (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-01-25; First posted 2011-01-31 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Colorectal Carcinoma
Keywords: Colon Cancer; Rectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Ramucirumab; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFIRI plus Ramucirumab (IMC-1121B) (Experimental)
  Interventions: Biological: Ramucirumab (IMC-1121B); Drug: Irinotecan; Drug: levofolinate; Drug: 5-Fluorouracil (5-FU)

INTERVENTIONS:
Biological: Ramucirumab (IMC-1121B) — Ramucirumab (IMC-1121B): Intravenous (IV) infusions, 8 milligrams per kilogram (mg/kg) every 2 weeks
  Other Names: IMC-1121B; Ramucirumab; LY3009806
Drug: Irinotecan — IV Infusion, 180 milligrams per square meter (mg/m²) every 2 weeks
Drug: levofolinate — IV infusion, 200 mg/m² every 2 weeks
Drug: 5-Fluorouracil (5-FU) — 400 mg/m² bolus followed by a 2400 mg/m² continuous infusion, every 2 weeks

SUMMARY:
The primary objective of this study is to investigate the safety and tolerability of the anti-vascular endothelial growth factor receptor-2 (anti-VEGFR-2) monoclonal antibody Ramucirumab (IMC-1121B) in combination with irinotecan, levofolinate, and 5-fluorouracil (FOLFIRI) in Japanese participants with advanced colorectal carcinoma (CRC).

ELIGIBILITY:
Inclusion Criteria:

* Participant is Japanese
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Has histologically or cytologically confirmed CRC
* Has metastatic disease that is not amenable to potentially curative resection
* Has received no more than 2 prior systemic chemotherapy regimens in any setting (only 1 prior regimen for metastatic disease is permitted)
* Has received first-line combination therapy of bevacizumab, oxaliplatin, and a fluoropyrimidine for metastatic disease and has experienced disease progression during first-line therapy, or disease progression within 6 months after the last dose of first-line therapy, or discontinued part or all of first-line therapy due to toxicity and experienced disease progression within 6 months after the last dose of first-line therapy. Participants must have received a minimum of 2 doses of bevacizumab as part of a first-line regimen containing chemotherapy in order to enroll.
* Has adequate hepatic, renal, hematologic, and coagulation function
* The participant's urinary protein is ≤1+ on dipstick or routine urinalysis. If urine dipstick or routine analysis indicates proteinuria ≥2+, then a 24-hour urine must be collected and must demonstrate <1000 milligrams (mg) of protein in 24 hours to allow participation in the study

Exclusion Criteria:

* Has received bevacizumab within 28 days prior to study registration
* Has received chemotherapy within 21 days prior to study registration
* Has received any previous systemic therapy (other than a combination of bevacizumab, oxaliplatin, and a fluoropyrimidine) for first-line treatment of metastatic CRC
* The participant experienced any of the following during first-line therapy with a bevacizumab-containing regimen: an arterial thrombotic/thromboembolic event; Grade 4 hypertension; Grade 4 proteinuria; a Grade 3-4 bleeding event; or bowel perforation
* Has received wide-field (full-dose pelvic) radiotherapy within 28 days prior to study registration
* Has undergone major surgery within 28 days or subcutaneous venous access device placement within 7 days prior to study registration
* Has elective or planned surgery to be conducted during the trial
* Has a history of deep vein thrombosis or pulmonary embolism within the past 12 months
* Has experienced any arterial thrombotic event within the past 12 months
* Participant is receiving therapeutic anticoagulation with warfarin, low-molecular weight heparin, or similar agents
* Participant is receiving chronic therapy with nonsteroidal anti-inflammatory agents [Aspirin up to 325 milligrams per day (mg/day) permitted]
* Has a significant bleeding disorder or has had a significant (Grade 3 or higher) bleeding event within 3 months prior to registration date
* Has a history of gastrointestinal perforation and/or fistulae within 6 months prior to registration date
* Has symptomatic congestive heart failure, unstable angina pectoris, or symptomatic or poorly controlled cardiac arrhythmia
* Has uncontrolled arterial hypertension despite standard medical management
* Has a serious or nonhealing wound, peptic ulcer, or bone fracture within 28 days prior to study registration
* Has an acute/subacute bowel obstruction or history of clinically significant chronic diarrhea
* Has a history of inflammatory bowel disease or Crohn's disease requiring medical intervention within 12 months prior to registration date
* The participant has either peptic ulcer disease associated with a bleeding event or known active diverticulitis
* Has an active infection requiring antibiotic, antifungal, or antiviral therapy
* Has known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related illness
* Has known leptomeningeal or brain metastases or uncontrolled spinal cord compression
* Has a known history of Gilbert's Syndrome, or is known to have any of the following genotypes: uridine diphosphate glucuronosyltransferase 1 family, polypeptide A1 (UGT1A1)*6/*6; UGT1A1*28/*28 or UGT1A1*6/*28
* Has previous or concurrent malignancy, except for basal or squamous cell skin cancer and/or in situ carcinoma, or other solid tumors treated curatively and without evidence of recurrence for at least 3 years

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Japan (3):
  - ImClone Investigational Site, Chiba
  - ImClone Investigational Site, Osaka
  - ImClone Investigational Site, Shizuoka

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eight (8) participants signed the informed consent.
Groups:
- FOLFIRI Plus Ramucirumab (IMC-1121B): Ramucirumab (IMC-1121B): Intravenous (IV) infusion, 8 milligrams per kilogram (mg/kg) every 2 weeks. Then 1-hour observation followed by chemotherapy with irinotecan, levofolinate, and 5-fluorouracil (FOLFIRI) according to manufacturer's standards. Irinotecan: IV infusion, 180 milligrams per square meter (mg/m^2) every 2 weeks. Levofolinate: IV infusion, 200 mg/m^2 every 2 weeks. 5-fluorouracil (5-FU): 400 mg/m^2 bolus followed by a 2400 mg/m^2 continuous infusion, every 2 weeks.
  Antiemetic premedication recommended according to manufacturer's standards but not required prior to ramucirumab drug product infusion. Participants who did not experience unacceptable toxicities during dose limiting toxicity (DLT) assessment period (Day 1, Cycle 1 through Day 1, Cycle 3) who met criteria for treatment continuation received additional cycles of study medication until disease progression, unacceptable toxicity, protocol noncompliance, withdrawal of consent, or Sponsor/investigator decision.
Period: Overall Study
Arm/Group | FOLFIRI Plus Ramucirumab (IMC-1121B)
Started | 6
Completed DLT Assessment Period | 5
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety population: Participants who received any quantity of study medication.
Arm/Group | FOLFIRI Plus Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 6
Region of Enrollment [Number; unit: participants]
  Japan | 6
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — ECOG performance status classified participants according to their functional impairment. Scores ranged from 0 (fully active) to 5 (death).
  participants
    0 - Fully active | 3
    1 - Ambulatory, restricted strenuous activity | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experienced Any Dose-Limiting Toxicities (DLT) During the DLT Assessment Period
Description: DLTs were adverse events (AEs) possibly related to study drug that met the National Cancer Institute's Common Terminology Criteria for AEs (NCI CTCAE, version 4.03): Grade 4 neutropenia ≥7 days or ≥Grade 3 with bacteremia or sepsis; Absolute neutrophil count <1.0x10^9/Liters with fever ≥38.3°Celsius requiring intravenous antibiotic therapy; Grade 4 thrombocytopenia or ≥Grade 3 with bleeding requiring platelet transfusion; ≥Grade 3 altered coagulation tests and no anticoagulation; ≥Grade 4 or uncontrolled hypertension; ≥Grade 3 non-hematologic toxicity (except non-clinically significant Grade 3 events like electrolyte abnormality, hypersensitivity, and arthralgia/myalgia); urine protein >3 grams/24 hours; study drug-related toxicity causing Cycle 3, Day 1 treatment delay until Day 44 or later. Grade 3 or Grade 4 infusion-related reaction (hypersensitivity) due to ramucirumab or FOLFIRI, not a DLT.
Time Frame: Day 1, Cycle 1 through Day 1, Cycle 3 (1 cycle=14 days)
Population: DLT population: All enrolled participants who either completed the first 3 administrations of study medication or discontinued study medication due to a DLT during the DLT assessment period (Day 1, Cycle 1 through Day 1, Cycle 3).
Measure: Number; unit: participants
Arm/Group | FOLFIRI Plus Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 6
participants | 1

2. Primary Outcome: Number of Participants With Ramucirumab Drug-Related Adverse Events or Serious Adverse Events
Description: Data are presented for the number of participants who experienced treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), Grade ≥3 TEAEs, or adverse events (AEs) leading to discontinuation of treatment that were considered to be related to ramucirumab. Events related to Irinotecan, Levofolinate, and 5-fluorouracil (5-FU) were reported separately. A summary of SAEs and other nonserious AEs, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline to end of study (up to 49.3 weeks) plus 37 day follow-up
Population: Safety population: Participants who received any quantity of study medication.
Measure: Number; unit: participants
Arm/Group | FOLFIRI Plus Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 6
participants
  Related TEAE | 6
  Related SAE | 0
  Related Grade ≥3 TEAE | 3
  Related AE leading to discontinuation | 2

3. Secondary Outcome: Number of Participants With Serum Anti-IMC-1121B Antibodies (Immunogenicity)
Time Frame: Day 1 of Cycle 5 (Week 9), Cycle 6 (Week 11), Cycle 7 (Week 13), and Cycle 9 (Week 17) [(1 cycle=14 days)]
Population: Participants who received any quantity of study medication and had evaluable immunogenicity data at the specified time points.
Measure: Number; unit: participants
Arm/Group | FOLFIRI Plus Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 5
participants
  Day 1, Cycle 5 (n=5) | 0
  Day 1, Cycle 6 (n=1) | 0
  Day 1, Cycle 7 (n=3) | 0
  Day 1, Cycle 9 (n=4) | 0

4. Secondary Outcome: Maximum Concentration (Cmax) of Ramucirumab
Description: The Cmax of ramucirumab in serum on Day 1, Cycle 1 and on Day 1, Cycle 5, which was also considered Cmax at steady state (Cmax,ss), is reported.
Time Frame: Day 1, Cycle 1 and Day 1, Cycle 5 (1 cycle=14 days)
Population: Participants who received any quantity of study medication and had evaluable Cmax data at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | FOLFIRI Plus Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 6
micrograms per milliliter (mcg/mL)
  Day 1, Cycle 1 (n=6) | 245 (6)
  Day 1, Cycle 5 (n=2) | 267 (11)

5. Secondary Outcome: Area Under the Curve (AUC) of Ramucirumab
Description: Reported for Day 1, Cycle 1 is AUC from time 0 extrapolated to infinity [AUC(0-inf)] and for Day 1, Cycle 5 is AUC over the dosing interval at steady state AUC(tau,ss).
Time Frame: Day 1, Cycle 1 and Day 1, Cycle 5 (1 cycle=14 days)
Population: Participants who received any quantity of study medication and had evaluable AUC data at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*day/milliliter (mcg*day/mL)
Arm/Group | FOLFIRI Plus Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 4
micrograms*day/milliliter (mcg*day/mL)
  Day 1, Cycle 1 (n=4) | 1600 (15)
  Day 1, Cycle 5 (n=2) | 1690 (38)

6. Secondary Outcome: Half Life (t1/2) of Ramucirumab
Description: t1/2 is the time required for the plasma/serum concentration to decrease 50%.
Time Frame: Day 1, Cycle 1 and Day 1, Cycle 5 (1 cycle=14 days)
Population: Participants who received any quantity of study medication and had evaluable t1/2 data at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | FOLFIRI Plus Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 6
days
  Day 1, Cycle 1 (n=6) | 7.38 (19)
  Day 1, Cycle 5 (n=2) | 8.55 (2)

7. Secondary Outcome: Clearance (CL) of Ramucirumab
Description: The total body CL of ramucirumab on Day 1, Cycle 1 and on Day 1, Cycle 5, which was also considered CL at steady state (CLss), is reported.
Time Frame: Day 1, Cycle 1 and Day 1, Cycle 5 (1 cycle=14 days)
Population: Participants who received any quantity of study medication and had evaluable CL data at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters per hour (mL/hr)
Arm/Group | FOLFIRI Plus Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 4
milliliters per hour (mL/hr)
  Day 1, Cycle 1 (n=4) | 11.4 (26)
  Day 1, Cycle 5 (n=2) | 10.4 (61)

8. Secondary Outcome: Steady State Volume of Distribution (Vss) of Ramucirumab
Description: Vss is the theoretical volume in which the total amount of study drug would need to be uniformly distributed during steady state to produce the same concentration as it is in plasma/serum.
Time Frame: Day 1, Cycle 1 and Day 1, Cycle 5 (1 cycle=14 days)
Population: Participants who received any quantity of study medication and had evaluable Vss data at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | FOLFIRI Plus Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 4
Liters (L)
  Day 1, Cycle 1 (n=4) | 2.51 (25)
  Day 1, Cycle 5 (n=2) | 3.06 (56)

9. Secondary Outcome: Best Overall Response [Anti-Tumor Activity of FOLFIRI Plus Ramucirumab (IMC-1121B)]
Description: Best overall response evaluated using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1) criteria. Complete Response (CR): disappearance of all non-nodal target lesions, with the short axes of any target lymph nodes reduced to <10 millimeters (mm). Partial Response (PR): at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph nodes), taking as reference the baseline sum diameter. Progressive Disease (PD): an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum on study (included baseline sum if that was the smallest on study). In addition, the sum must have demonstrated an absolute increase of at least 5 mm (the appearance of 1 or more new lesions was considered progression). Stable Disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD, taking as reference the smallest sum diameter since treatment started.
Time Frame: Every 8 weeks until PD (up to 49 weeks)
Population: Safety population: Participants who received any quantity of study medication.
Measure: Number; unit: participants
Arm/Group | FOLFIRI Plus Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 6
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 1
  Stable Disease (SD) | 4
  Progressive Disease (PD) | 1

ADVERSE EVENTS:
Arm/Group | FOLFIRI Plus Ramucirumab (IMC-1121B)
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | FOLFIRI Plus Ramucirumab (IMC-1121B) (N=6)
ANAEMIA (Blood and lymphatic system disorders) | 1 (3)
NEUTROPENIA (Blood and lymphatic system disorders) | 5 (34)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (11)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (3)
CHEILITIS (Gastrointestinal disorders) | 1 (2)
DIARRHOEA (Gastrointestinal disorders) | 5 (12)
GINGIVITIS (Gastrointestinal disorders) | 1 (1)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (3)
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 3 (34)
PERIODONTAL DISEASE (Gastrointestinal disorders) | 2 (2)
STOMATITIS (Gastrointestinal disorders) | 5 (12)
VOMITING (Gastrointestinal disorders) | 4 (22)
FACE OEDEMA (General disorders) | 1 (1)
FATIGUE (General disorders) | 3 (5)
FEELING ABNORMAL (General disorders) | 1 (1)
INFUSION RELATED REACTION (General disorders) | 1 (1)
MALAISE (General disorders) | 2 (23)
OEDEMA (General disorders) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 2 (4)
NASOPHARYNGITIS (Infections and infestations) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (2)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
SKIN INJURY (Injury, poisoning and procedural complications) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1)
WEIGHT DECREASED (Investigations) | 1 (2)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (3)
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 (36)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (2)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 (3)
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 1 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 1 (2)
INSOMNIA (Psychiatric disorders) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 2 (10)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1/2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (6)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (2)
HYPERTENSION (Vascular disorders) | 1 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.